CLINICAL TRIAL: NCT06672731
Title: BIODETECT_CP a Novel Combination of BIOchemical, DEnsitometric, TEChnological and Imaging Tools to Evaluate the Bone/muscle Unit Health in Children with Cerebral Palsy
Brief Title: BIOchemical, DEnsitometric, TEChnological and Imaging Tools to Evaluate the Bone/muscle in Children with Cerebral Palsy
Acronym: BIODETECT_CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: University of Pisa (Other); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRIN2022; PRIN2002 (Other Grant/Funding Number: Italian Ministry of Education)
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy Infantile
Keywords: cerebral palsy; bone health; muscle health
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Children with cerebral palsy (Experimental): 50 children with cerebral palsy in whom the intervention is intended as the application of already validated movement sensors, namely actigraphs.
  Interventions: Diagnostic Test: REMS: Radiofrequency Echographic Multi Spectrometry
- Typically developing children (Active Comparator): 50 healthy children, evaluated c/o AOUP for the exclusion of other diseases, in whom for intervention is intended the application of already validated movement sensors.
  Interventions: Diagnostic Test: REMS: Radiofrequency Echographic Multi Spectrometry

INTERVENTIONS:
Diagnostic Test: REMS: Radiofrequency Echographic Multi Spectrometry — it is a non invasive ultrasonographic evaluation of bone and muscle quality

SUMMARY:
Cerebral palsy (CP) is the most common chronic disability in childhood, burden by motor, sensation, cognition, feeding and communication impairment. A serious concern in children with CP is bone/muscle health deterioration, which negatively impacts the already reduced quality of life (QoL). Children with CP show low bone density, vitamin D deficiency, sarcopenia and high risk of fragility fractures, with heavy effects on what is already limited home, school and community life. The causes for muscle-bone impairment are low weight-bearing deambulation during skeletal formation with low bone mineralization, poor nutrition and low calcium intake, low sun exposure, use of anticonvulsant medications with a negative profile on bone. Understanding the causes affecting bone quality and setting up interventions to reduce the impact of physical disability are essential in young subjects with CP.

This project combines complementary expertise and resources in the fields of Endocrinological Biochemistry, Paediatric Neurological Disorders and Neuroimaging, to allow an innovative, technology-assisted workup for bone/muscle health evaluation in young subjects with CP, which could drive novel therapeutics, nutritional and rehabilitation programs.

The first aim of this project is to evaluate bone/muscle health in young subjects with CP compared with sex-age matched healthy subjects, providing i) serum biomarkers of mineral metabolism and the metabolome of Vitamin D, assessed with last generation Mass Spectrometry, ii) muscle sarcopenia markers like Irisin and other myokines, depicting the response of the muscle to exercise iii) neuronal damage and inflammatory markers, iv) densitometric data by the low-cost and safe Quantitative ultrasound (QUS) at phalanges of the hand, plus the novel and very promising Radiofrequency Echographic Multi Spectrometry (REMS) served by the software for fragility fractures risk.

We also aim to correlate the previous mentioned markers of bone/muscle health with a combination of demographic, clinical, cognitive and technological parameters, the last obtained by an innovative use of wearable sensors or actigraphs, positioned at the wrists, which depicts movements, physical activity (PA), energy expenditures (EE) and, together with heart-rate monitors, metabolic data during a normal like week in subjects with CP and healthy controls. Finally, a newly validated scoring for brain lesions in subjects with CP and the production of imaging "biomarkers" of neuronal damage, will be correlated with their bone/muscle health data, PA and EE to understand the impact of brain damage on functional performance and bone metabolism.

DETAILED DESCRIPTION:
This study investigates the correlation between brain lesions, physical ability, and bone/muscle health in young patients with cerebral palsy (CP). It posits that:

Bone and muscle health in young individuals with CP is compromised, affecting their quality of life and development. The study aims to utilize biomarkers related to bone fragility, sarcopenia, and neuronal damage, alongside advanced imaging techniques (quantitative ultrasound and Radiofrequency Echographic Multi Spectrometry) to assess bone/muscle unit health accurately.

Physical activity limitations and reduced energy expenditure negatively impact bone/muscle health in CP patients. The researchers plan to leverage wearable sensors to provide precise measurements of physical activity and correlate these with the established biomarkers and imaging results, aiding in customized treatment approaches.

Brain MR imaging could reveal structural changes in the brain, which may correlate with physical activity and bone/muscle health data, helping to understand the implications of brain damage on overall functionality.

The objectives include comparing bone/muscle health between children with CP and healthy peers, assessing physical activity's impact on bone/muscle health, and analyzing brain imaging results in relation to those health metrics. The study anticipates enrolling 50 participants with CP and 50 age-matched controls, utilizing various biochemical and imaging techniques to gather and compare data on bone and muscle health, physical activity, and brain lesions.

ELIGIBILITY:
Inclusion Criteria:

* age
* willing to sign inform content

Exclusion Criteria:

* bisphosphonates or bone diseases

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone/Muscle Unit Health Assessment | at enrollment
  We will achieve the aim 1 by the following evaluations:
  - 25OHD changes evaluated as plasma levels of Vitamin D, intended as hypovitaminosis D 25OHD<20 ng/ml
Evaluation of bone mineral density as QUS | at enrollment
  AD-SOS (amplitude-dependent speed of sound) expressed as standard deviation compared to normal (absolute number) and BTT (bone transmission time expressed in seconds)
Evaluation of bone/muscle score at REMS | at enrollment
  T score and Z score at REMS are index of bone fagility and are expressed as standard deviation difference compared to normal (absolute number, cut off <2.5). Moreover a % of fragility risk is produced (cut-off >10%)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tinelli F, Guzzetta A, Purpura G, Pasquariello R, Cioni G, Fiori S. Structural brain damage and visual disorders in children with cerebral palsy due to periventricular leukomalacia. Neuroimage Clin. 2020;28:102430. doi: 10.1016/j.nicl.2020.102430. Epub 2020 Sep 11. PMID 32980597
- [Background] Di Paola M, Gatti D, Viapiana O, Cianferotti L, Cavalli L, Caffarelli C, Conversano F, Quarta E, Pisani P, Girasole G, Giusti A, Manfredini M, Arioli G, Matucci-Cerinic M, Bianchi G, Nuti R, Gonnelli S, Brandi ML, Muratore M, Rossini M. Radiofrequency echographic multispectrometry compared with dual X-ray absorptiometry for osteoporosis diagnosis on lumbar spine and femoral neck. Osteoporos Int. 2019 Feb;30(2):391-402. doi: 10.1007/s00198-018-4686-3. Epub 2018 Sep 4. PMID 30178159
- [Background] Tomai Pitinca MD, Fortini P, Gonnelli S, Caffarelli C. Could Radiofrequency Echographic Multi-Spectrometry (REMS) Overcome the Limitations of BMD by DXA Related to Artifacts? A Series of 3 Cases. J Ultrasound Med. 2021 Dec;40(12):2773-2777. doi: 10.1002/jum.15665. Epub 2021 Feb 21. PMID 33615539
- [Background] Baroncelli GI. Quantitative ultrasound methods to assess bone mineral status in children: technical characteristics, performance, and clinical application. Pediatr Res. 2008 Mar;63(3):220-8. doi: 10.1203/PDR.0b013e318163a286. PMID 18287958
- [Background] Colaianni G, Faienza MF, Sanesi L, Brunetti G, Pignataro P, Lippo L, Bortolotti S, Storlino G, Piacente L, D'Amato G, Colucci S, Grano M. Irisin serum levels are positively correlated with bone mineral status in a population of healthy children. Pediatr Res. 2019 Mar;85(4):484-488. doi: 10.1038/s41390-019-0278-y. Epub 2019 Jan 15. PMID 30683930
- [Background] Saggese G, Vierucci F, Prodam F, Cardinale F, Cetin I, Chiappini E, De' Angelis GL, Massari M, Miraglia Del Giudice E, Miraglia Del Giudice M, Peroni D, Terracciano L, Agostiniani R, Careddu D, Ghiglioni DG, Bona G, Di Mauro G, Corsello G. Vitamin D in pediatric age: consensus of the Italian Pediatric Society and the Italian Society of Preventive and Social Pediatrics, jointly with the Italian Federation of Pediatricians. Ital J Pediatr. 2018 May 8;44(1):51. doi: 10.1186/s13052-018-0488-7. PMID 29739471
- [Background] Braito I, Maselli M, Sgandurra G, Inguaggiato E, Beani E, Cecchi F, Cioni G, Boyd R. Assessment of upper limb use in children with typical development and neurodevelopmental disorders by inertial sensors: a systematic review. J Neuroeng Rehabil. 2018 Nov 6;15(1):94. doi: 10.1186/s12984-018-0447-y. PMID 30400992